CLINICAL TRIAL: NCT06159946
Title: Access-H20: Sensor Driven Smart Faucet to Enable and Empower Independent Drinking and Grooming for Individuals Impacted by Spinal Cord Injury
Brief Title: Access-H20 Faucet for Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Old Dominion University (Other)
Responsible Party: Principal Investigator, Anna Jeng, Professor, Old Dominion University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 1R43HD108061-01A1 (NIH)
Record Dates: First submitted 2023-10-04; First posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Spinal Cord Injury Cervical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spinal cord injury (Experimental): Each subject was asked to place their hand by the motion sensor (motion control), use a speech speaker (voice control), and then move their eyes up, down, left, and right to activate the eye gaze sensor (eye gaze control) to control water outputs for drinking, rinsing, and grooming. Each subject performed the same task/function three times.
  Interventions: Device: Access-H2O faucet

INTERVENTIONS:
Device: Access-H2O faucet — The assigned invention was developed to test the feasibility of the prototype of the Access-H2O faucet by assessing whether subjects can activate the faucet to control water outputs via the motion sensor, eye gaze, and a speech speaker. To activate the faucet via the motion sensor, each subject was asked to place his or her hand near the motion sensor. To activate the faucet via the eye gaze, each subject was asked to look directly at the eye gaze sensor. To activate the faucet via the speech speaker, each subject was asked to speak to the speaker. Each subject performed the same function three times. The water from the faucet was used for drinking, rinsing, and grooming.

SUMMARY:
The Phase I SBIR objective is to design, develop & demonstrate feasibility of Access-H2OTM, a sensor driven smart faucet to enable and empower independent drinking and grooming for individuals impacted by spinal cord injury (SCI). SCI severely impacts functional independence & ability to perform activities of daily living (ADLs). Greater function is typically lost with higher, more complete injuries. More specifically, those impacted above C5-C7 have impaired upper extremities, which limits the use of arms and hands for activities such as eating, drinking, and grooming. Functional access to water for these individuals becomes a key to increased independence and successful completion of ADLs. Therefore, commercialization of smart fountain faucets, which can automatically deliver water in target temperature, force, & nozzle setting for a specific ADL, has the potential to empower individuals with SCI for greater independence & and improved quality of life. Subjects with SCI and controls were recruited to test the functionality of the faucet which includes eye gaze, voice, and motion sensors to control the water stream for drinking, rinsing, and grooming.

DETAILED DESCRIPTION:
Nearly 300,000 individuals are living with spinal cord injuries (SCI), and over 12,000 new SCI occur annually in the United States. Most SCIs involve the cervical (neck) region of the spine and cause partial or complete loss of movement of both arms, both legs, and the torso (quadriplegia). Individuals with a higher-level and more complete SCI typically have greater loss of functional movement and sensation below the level of the injury. They require greater levels of assistance for self-care and mobility. Currently, there are limited options for quadriplegics to access water to perform basic activities of daily living such as drinking. Additionally, hydration packs and straws create unsanitary conditions and can be difficult to use. The aim of the project is to develop an innovative fountain faucet to enable individuals living with SCI to access water more independently for basic activities of daily living. The faucet incorporates electromechanical controls and software programs that adjust spray outlets, spray angles, and water temperatures. A proximity sensor and voice recognition function allow users to control the faucet through a smart speaker. These features enable precise dispensing of water at the desired temperature and volume, while a camera and other sensors enable hands-free operation. Subjects, including individuals living with SCI and controls, were recruited from an outpatient rehabilitation clinic to test the functionality of the faucet including eye gaze, voice, and motion sensors to control the water stream for drinking, rinsing, and grooming. The examiner screened the subjects to determine their levels of functional independence (independent, modified independent, assistance required, and dependent). The participants were also interviewed regarding their current methods of drinking, rinsing, and grooming. The percentage and standard deviation of individuals in each level of independence for each function were calculated. A t-test was conducted to determine any significant differences in the dependence levels between the tested subjects and the control group.

ELIGIBILITY:
Inclusion Criteria:

* Quadriplegics with injuries above C7

Exclusion Criteria:

* Subjects with cognitive deficits, serious mental health or medical conditions that would compromise subject safety or accurate user feedback will be excluded

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Water Access for Activities of Daily Living | The duration of time of assessment of the participant lasted for 2 to 3 hours.
  Each subject could complete the tasks: 1) Can the test participants get the water from the fountain faucet to their mouth to hydrate? 2) Can the test participants use the fountain feature to rinse their mouths? and 3) Can the test participants use the fountain spray to rinse a quarter-size area of soap partially or fully from their left and/or right cheeks? Coding 1 was labeled as "successful," coding 2 as "partially successful," and coding 3 as "not completed." A System Usability Scale was determined.

CONTACTS AND LOCATIONS:
Locations (1):
- ODU Monarch Physical Therapy Clinic, Norfolk, Virginia, United States

DOCUMENTS (1):
  • Study Protocol (2022-03-22): https://cdn.clinicaltrials.gov/large-docs/46/NCT06159946/Prot_000.pdf